CLINICAL TRIAL: NCT05735379
Title: Impact in Older Adults of Reducing Anticholinergic and Sedative Medication Burden on Physical Function Measured by Clinical Digital Phenotyping in Lab and Real-life Environments
Brief Title: Impact in Older Adults of Reducing Anticholinergic and Sedative Rx Burden on Physical Function Measured by Wearables
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de recherche du Centre hospitalier universitaire de Sherbrooke (Other)
Responsible Party: Principal Investigator, Benoit Cossette, Professor, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PJT-183968
Record Dates: First submitted 2023-01-26; First posted 2023-02-21 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Deprescribing Anticholinergic and Sedative Medications; Physical Function
MeSH Terms: interventions — Drug Tapering

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deprescribing anticholinergic and sedative medications (Experimental): Deprescribing plan targeting a reduction in drug burden index score of ≥ 0.5
  Interventions: Drug: Deprescribing anticholinergic and sedative mediications

INTERVENTIONS:
Drug: Deprescribing anticholinergic and sedative mediications — Deprescribing plan targeting a reduction in Drug Burden Index score of ≥ 0.5
  Other Names: Drug cessation or dose reduction

SUMMARY:
Medications with sedative or anticholinergic effects such as antidepressants, benzodiazepines, or opioids have been associated with impaired cognitive and physical function. They are referred to as potentially inappropriate medications or medications that are best avoided by older adults. The accumulated evidence has now shifted the clinical and research focus to evaluating the who, what, and how of the best way to deprescribe (i.e., dose reduction or cessation of these medications). The Drug Burden Index (DBI) allows researchers and clinicians to quantify the cumulative burden of anticholinergic and sedative medications in each patient. Deprescribing these medications is a complex health intervention based on trade-offs between their clinical benefits (e.g., symptom management and prevention of diseases) and their adverse drug events to improve physical and cognitive function. Existing physical function performance metrics, such as gait speed captured in the clinic, are often non-specific and do not reflect real-life performance. Innovative mobility metrics are required to better understand specific deficits with age and disease and the effects of medications on these deficits.

The goal of this project is to better characterize the impact of reducing the anticholinergic and sedative medication burden on physical function in older adults by novel mobility metrics in lab and real-life environments.

A prospective, longitudinal cohort of 182 community-dwelling older adults (≥ 65 years) with a DBI of ≥ 1 will be completed. Using a quasi-experimental design, recruited patients will undergo a medication deprescribing plan, as part of usual clinical care, that includes three gradual changes to their medication regimen resulting in three DBI levels. At each DBI level, physical function mobility including dual-task tests) will be assessed in the lab with wearable sensors during validated clinical tests such as the Short Physical Performance Battery. Objective balance and mobility metrics (e.g., sway area and frequency, stride length) will be extracted. Physical function will also be assessed continuously in the patient's real-life environment from recruitment to the last lab visit, using wearable (Apple Watch® with ankle inertial measurement unit) and environmental sensors. Cognition will be measured using the Montreal Cognitive Assessment, Trail Making Test Part A & B, and Digit Symbol Substitution Test.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and older
* community-dwelling
* Drug Burden Index score of ≥ 1
* Agree with a deprescribing plan targeting a reduction in Drug Burden Index score of ≥ 0.5.

Exclusion Criteria:

* Dementia
* Need of a walker as a mobility assistive device
* Unstable medical condition (≥ 1 unplanned hospitalization or ≥ 2 emergency department visits in the past month).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in gait capacity measured in the lab from baseline to study completion | Through study completion, an average of 4 months.
  Gait speed (m/s)

SECONDARY OUTCOMES:
Change in gait performance measured in real-life settings from baseline to study completion | Through study completion, an average of 4 months.
  Gait activity (number of steps)
Change in functional limitations and disability from baseline to study completion | Through study completion, an average of 4 months.
  Late-Life Function and Disability Instrument (Late-Life FDI),
Change in caregiver report of the patients' functional status from baseline to study completion | Through study completion, an average of 4 months.
  Older Adults Resources and Services (OARS) Multidimensional Functional Assessment Questionnaire adapted for the caregiver.
Change in falls and near falls from baseline to study completion | Through study completion, an average of 4 months.
  Falls nand near falls recorded by patient diary
Change in falls and near falls from baseline to study completion | Through study completion, an average of 4 months.
  Falls and near falls recorded from the Apple Watch® proprietary algorithm.
Adverse drug events and adverse drug withdrawal events | Continuous during the deprescribing process
  Adverse anticholinergic and sedative effects from G-MEDSS
Change in Montreal Cognitive Assessment (MoCA) from baseline to study completion | Through study completion, an average of 4 months.
  Full version
Change in Trail Making Test (TMT) from baseline to study completion | Through study completion, an average of 4 months.
  Part A & B
Change in Digit Symbol Substitution Test from baseline to study completion | Through study completion, an average of 4 months.
  DSST

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided